CLINICAL TRIAL: NCT06466356
Title: Psychoeducational Course for Suicide Prevention - a Randomized Controlled Trial
Brief Title: Psychoeducational Course for Suicide Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Helse Nord-Trøndelag HF (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 142708
Record Dates: First submitted 2024-06-03; First posted 2024-06-20 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Suicide Prevention; Suicide Threat; Self Efficacy; Stress, Psychological; Psychiatric Emergency; Psychiatric Disorder
Keywords: Psychoeducation; Safety plan; Gatekeeper; Suicidal crisis syndrome
MeSH Terms: conditions — Suicide Prevention; Stress, Psychological; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients acutely admitted to Department of acute psychiatry, St Olav University Hospital (SOH) or Levanger Hospital or acutely admitted to an outpatient team for acute and emergency psychiatry, SOH, or admitted to a district psychiatric centers (DPS) in Trøndelag county or evaluated by physicians or psychologists at the Consultation Liaison, SOH. Patients will be included with consecutive sampling of patients who meet the selection criteria and give an informed consent.
  Participants will be equally randomized (1:1) in the intervention and control group and randomization will take place by digital randomization using WebCRF (KlinForsk/ Klinisk forskningsenhet Midt-Norge). Stratified randomization will be used regarding the baseline variable "substance abuse", ensuring that this variable is more evenly distributed between the two groups than chance.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patient and treating clinician will be unblinded to treatment modality. To compensate for lack of blinding concerning the received treatment, the persons ratings, subsequent measurements and data collection at follow-up will be blinded to the treatment conditions to avoid confirmation bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducational group therapy (Experimental): Group therapy session, 3 meetings. Each group includes 8-10 participant to receive a group based psychoeducative intervention (three for patients, one for next of kin) and TAU.
  Interventions: Other: Psychoeducational Course for Suicide Prevention; Other: Treatment as usual
- Individual therapy session (Active Comparator): The participants in the control group receive one individual therapy session with focus on suicide risk and safety plan with a psychologist or physician and TAU
  Interventions: Other: Individual therapy session; Other: Treatment as usual

INTERVENTIONS:
Other: Psychoeducational Course for Suicide Prevention — Baseline variables includes diagnosis using ICD-10 criteria for research and demographic variables such as age, sex, level of education and occupation. Following assessments will be used when including patients for the project: The General self-efficacy scale (GSE) with additional questions related to the theme of the psychoeducational topics, The mental pain questionnaire (MPQ, Alcohol Use Disorders Identification Test (AUDIT), Drug Use Disorders Identification Test (DUDIT) The Patient Health Questionnaire (PHQ-9), GAD-7, The SCS-Checklist and SCI-5. GSE, MPQ and PHQ-9 will be measured after intervention and after 6, 12, 24 and 60 months.
  Arms: Psychoeducational group therapy
Other: Individual therapy session — Baseline variables includes diagnosis using ICD-10 criteria for research and demographic variables such as age, sex, level of education and occupation. Following assessments will be used when including patients for the project: The General self-efficacy scale (GSE) with additional questions related to the theme of the psychoeducational topics, The mental pain questionnaire (MPQ, Alcohol Use Disorders Identification Test (AUDIT), Drug Use Disorders Identification Test (DUDIT) The Patient Health Questionnaire (PHQ-9), GAD-7, The SCS-Checklist and SCI-5. GSE, MPQ and PHQ-9 will be measured after intervention and after 6, 12, 24 and 60 months.
  Arms: Individual therapy session
Other: Treatment as usual — Treatment as usual (TAU) may include the use of psychotropic drugs, in and out-patient treatment, occupational therapy and other interventions the patients physician deem necessary.

SUMMARY:
The plan is to include patients with a history of increased risk of suicide. In the aftermath of an episode of imminent suicide risk, patients will receive a psychoeducational course that entails information on different aspects of suicide-related topics, identifying triggers and detecting early warning signals for increased suicide risk. The course culminates in working on completing a individual safety plan to prevent an future increase in suicide risk. The course will incorporate both patients and their next of kin. The psychoeducational course will be compared to a control group where the patients receive one individual session with focus on a safety plan to evaluate the intervention. Both groups will receive treatment as usual (TAU) during both the acute phase and follow-up. The study will be conducted as a randomized controlled trial.

DETAILED DESCRIPTION:
Patients will be included during admittance in the acute psychiatric ward or when in contact with the outpatient team for acute and emergency psychiatry. They will receive acute treatment and be placed on a waiting list until enough patients are included to start the intervention. Then the included patients will be randomized to either the psychoeducational course or the individual session. The course and the individual lessons start at the same time. Each group includes 8-10 participant to receive a group based psychoeducative intervention (three for patients, one for next of kin) and TAU.

The first session (2x45 min) focus on information on suicidal thoughts, mental pain, suicide attempts and suicide as a phenomenon with focus on vulnerability factors, risk development and development of the suicidal crisis syndrome. The second session (2x45 min) tackles identifying triggers for increase in suicide risk and suicidal impulses, detecting early warning signals for increased suicide risk and how to recognize the change as it happens. In the third session (3x45 min) patients work on completing the individual safety plan to prevent an increase in suicide risk. The plan includes "situations that may trigger increased risk", "how to recognize and communicate the increased risk" and "actions that may reduce or increase risk." Finally, the fourth and last session (2x45 min) is aimed at the next of kin that the group participant wants to attend. Patients do not attend this session. The next of kin receive a review of the information from the first two sessions, as well as focus on what the next of kin can or cannot do to help if the risk of suicide increases.

The control group receive one individual session with focus on suicide risk and safety plan with a psychologist or physician and TAU.

Randomization and masking of study groups Participants will be equally randomized (1:1) in the intervention and control group. Patients will be included during admittance in the acute psychiatric ward or when in contact with the outpatient team for acute and emergency psychiatry. The first randomization takes place when sixteen to twenty participants are included. Randomization will take place by manual randomization by an external person at the Research department at St. Olav Hospital in Trondheim. This ensures an equal distribution between the intervention group and the control group. The patient and treating clinician will be unblinded to treatment modality. To compensate for lack of blinding concerning the received treatment, the persons ratings, subsequent measurements and data collection at follow-up will be blinded to the treatment conditions to avoid confirmation bias. The statistical advisor will also be blinded to treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suicide attempt, suicidal behavior, or risk of suicidal behavior and a clinician evaluating that the patient has an intention to die
* Patients with a suicide attempt or suicidal behavior defined as "a self-inflicted, potentially injurious behavior with a non-fatal outcome for which there is evidence of intention of death and/or considered to have had or been close to a suicidal crisis syndrome.

Exclusion Criteria:

* Not being sufficiently fluent in Norwegian to provide informed consent, valid responses on psychometric testing or to benefit from a psychoeducative course.
* A known diagnosis of ICD-10 F 60.3 (borderline personality disorder) with similar symptoms at previous admittances.
* Ongoing psychosis.
* A substance abuse condition to such a degree that they are unable to comply with the protocol and are considered to be at risk when attending psychoeducational courses.
* Organic brain disorders or mental disabilities in such a degree that they are unable to comply with the protocol.
* Not being able to give an informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Self efficacy | Immediately after completing the course/ individual sessions. Thereafter within one month after 6, 12, 24 and 60 months after completing the course/ individual sessions.
  The General self-efficacy scale (GSE) measures optimistic self-beliefs in coping with the demands, tasks and challenges of life in general. It consists of 10 statements that respondents rate on a scale from 1 (not at all true) to 4 (exactly true). The individual's scores on each item are summed up to a GSE score with higher scores indicating higher GSE. Questions regarding the perceived efficacy regarding handling future episodes of increased suicide is added. An increase of ≥ 5 points on the GSE scale is considered the limit for a minimally clinically important change.

SECONDARY OUTCOMES:
Mental pain | Immediately after completing the course/ individual sessions. Thereafter within one month after 6, 12, 24 and 60 months after completing the course/ individual sessions.
  The mental pain questionnaire (MPQ). The MPQ includes statements on sense of emptiness, loss of meaning and suffering. The statements are formulated on a dichotomous response format. Higher scores indicate higher level of mental pain. MPQ is a simple 10-items self-rating questionnaire and is a transdiagnostic tool. Minimum score 0, maximum score 10.
Symptoms of depression | Immediately after completing the course/ individual sessions. Thereafter within one month after 6, 12, 24 and 60 months after completing the course/ individual sessions.
  Symptoms measured by Patient Health Questionnaire (PHQ-9). The nine-item PHQ-9 is a depressive symptom scale. Scores range from minimum 0 to maximum 27. Higher scores indicate a worse outcome
Symptoms of anxiety | Immediately after completing the course/ individual sessions. Thereafter within one month after 6, 12, 24 and 60 months after completing the course/ individual sessions.
  The Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for screening and severity of anxiety. Scores range from minimum 0 to maximum 21. Higher scores indicate a worse outcome
Numbers of suicide attempts | At 6, 12, 24 and 60 months after the completion of the course/individual sessions.
  Suicide attempts recorded in the Norwegian Patient Registry (NPR).
Numbers of suicides | At 6, 12, 24 and 60 months after the completion of the course/individual sessions.
  Suicides recorded from the Norwegian Cause of Death Registry
Number of admittances in psychiatric hospital | At 6, 12, 24 and 60 months after the completion of the course/individual sessions.
  Admittances in psychiatric hospital recorded from Norwegian Patient Registry (NPR).
Number of days in psychiatric hospital | At 6, 12, 24 and 60 months after the completion of the course/individual sessions.
  Days in psychiatric hospital recorded from Norwegian Patient Registry (NPR).
Number of compulsory admissions | At 6, 12, 24 and 60 months after the completion of the course/individual sessions.
  Compulsory admissions recorded from Norwegian Patient Registry (NPR).
Number of voluntary admissions | At 6, 12, 24 and 60 months after the completion of the course/individual sessions.
  Voluntary admissions recorded from Norwegian Patient Registry (NPR).

CONTACTS AND LOCATIONS:
Overall Officials: Katrine K Fjukstad, PhD, Principal Investigator — Helse Nord Trøndelag
Locations (2):
- Norway (2):
  - Helse Nord-Trøndelag, Levanger, Trøndelag
  - St. Olav Hospital, Trondheim, Trøndelag

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT06466356/Prot_SAP_000.pdf